CLINICAL TRIAL: NCT00752154
Title: Curcumin in Rheumatoid Arthritis - ACross-Over Pilot Study
Brief Title: Curcumin in Rheumatoid Arthritis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 07-12-051
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2008-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Subjects; active; Rheumatoid; Arthritis; revised; American; College; Rheumatology; Criteria
MeSH Terms: conditions — Arthritis, Rheumatoid; Motor Activity; Arthritis | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Curcumin (Longvida™) — Curcumin (Longvida™) or matching placebo. They will begin by taking 4 capsules (approximately 2 grams) once a day for 2 weeks and then the dose will be increased to 4 capsules twice a day (4 gram per day) beginning at week 3. Subjects will remain at this dose for an additional 13 weeks for a total 16 weeks. After 16 weeks, the same procedures will be repeated for another 16 weeks

SUMMARY:
Curcuma longa or turmeric is a tropical plant native to south and southeast tropical Asia. Perhaps the most active component in turmeric is curcumin which may make up 2-5% of the total spice in turmeric. The study drug being tested in this study is curcumin.

This study is called a cross-over study because all subjects will receive the study drug for a certain amount of time and then switch to placebo (an inactive substance) for a certain time or vice versa. The subject's participation may last up to 8 months.

The subject will be randomized (by chance; like flipping a coin) to receive either the study drug, curcumin, or placebo for 4 months. After 4 months, if the subject was taking curcumin they will stop taking it and begin to take placebo and if the subject was taking placebo they will stop taking it and begin taking curcumin for the remaining 4 months. By completion of the study, all 40 subjects will have taken curcumin and placebo for 4 months each.

Curcumin/placebo will be provided in capsule form and the subject will take it by mouth. The dose dose will be increased every week for up to a total of 4 grams per day.

Subjects will have blood tests, complete questionnaires, and be seen by the study doctor.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years; read and understand English
2. Stable dose of non-steroidal anti-inflammatory agents (NSAID) for ≥ 2 weeks.
3. Oral prednisone or equivalent ≤ 10 mg daily and stable dose for ≥ 2 weeks(and must be kept stable throughout the duration of the protocol).

   * ESR > 20 mm/hr, or CRP > 0.8 mg/dl
4. May be using any of the following DMARDs: methotrexate, sulfasalazine, hydroxychloroquine or leflunomide. If using any of these DMARDs must be using them for ≥ 12 weeks and stable dose for ≥ 4 weeks. If using other DMARD, or DMARD combinations, these additional or other DMARDs must be stopped for ≥ 4 weeks before baseline visit. May also participate if patient not on DMARD,
5. Subjects must be diagnosed with rheumatoid arthritis based on the revised American College of Rheumatology criteria:Presence of > swollen and > 6 tender joint count (28 joint count), and either ESR > 20 mm/hr or CRP > 0.8 mg/dl

Exclusion Criteria:

1. Acute medical conditions deemed as inappropriate by the investigators (acute heart failure, uncontrolled diabetes mellitus, uncontrolled hypertension)
2. AST/ALT > 1.5 upper limit of normal (ULN)
3. Serum creatinine > 1.6 mg/dl
4. Hemoglobin/Hematocrit < 10.0 gram/dl/ 30.0
5. Platelet count < 100,000
6. Current use of warfarin (as there is a drug interaction between curcumin and warfarin).
7. Currently on biologic therapy (must have stopped etanercept for ≥ 4 weeks or adalimumab or infliximab for ≥ 8 weeks at time of Time 1 visit),
8. Women who are pregnant,
9. Subjects who are taking digoxin, warfarin and/or heparin,
10. Subjects with a history of antiphospholipid syndrome and other thrombophilic states,
11. Subjects who have an INR >= 1.5 at baseline,
12. Subjects with acute episode(s) of cholecystitis within the last 6 months,
13. Subjects with active peptic ulcer disease within the last 6 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2010-12-01 (Actual); Study Completion 2011-01-01 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology 20% | 4 month period

SECONDARY OUTCOMES:
Inflammatory cell signaling markers | 4 month
Safety of curcumin | 8 month

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Khanna, M.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Swamy Venuturpualli, M.D., 8737 Beverly Blvd., #203, Beverly Hills, California
  - UCLA, 1000 Veteran Avenue, Rehab Building, 3rd Floor, Los Angeles, California